CLINICAL TRIAL: NCT06839131
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase I Study to Evaluate Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of SPH9788 Tablet in Chinese Healthy Subjects.
Brief Title: A Clinical Study of SPH9788 Tablets in Healthy Chinese Subjects.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SPH9788-101
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-02

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPH9788 (Experimental)
  Interventions: Drug: SPH9788
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPH9788 — SPH9788 tablets administered orally
  Arms: SPH9788
Drug: Placebo — Matching placebo administered orally
  Arms: Placebo Comparator

SUMMARY:
The purpose of the study is to evaluate the safety of SPH9788 tablets in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects aged from 18 to 45 years;
2. Subject has a Body Mass Index (BMI) between 18.5 and 28.0 kg/m2 at screening and the weight of male subjects is not less than 50 kg, and the weight of female subjects is not less than 45 kg;;
3. Subjects who voluntarily participate and sign informed consent form;
4. Subjects who can communicate well with investigator and comply with the lifestyle restrictions specified in the protocol, and cooperate to complete the trial procedure;
5. Subjects willing to use reliable contraceptive methods throughout the trial and for 6 months after trial completion.

Exclusion Criteria:

1. Medical history (current or past) that in the investigator's judgment may interfere with trial participation;
2. Surgical/medical conditions that may significantly affect drug pharmacokinetics (absorption, distribution, metabolism, excretion) or pose safety risks;
3. Occurrence of protocol-defined exclusionary events within 3 months prior to investigational product administration;
4. Use of any prescription/non-prescription medications (including herbal products) within 2 weeks prior to dosing;
5. Known hypersensitivity to any component of the investigational product or history of severe allergic reactions;
6. Positive serology for hepatitis B surface antigen, hepatitis C antibody, HIV antibody, and syphilis serum reaction;
7. Substance abuse history within 1 year prior to screening or positive urine drug screen;
8. Alcohol abuse history within 1 year or positive alcohol breath test;
9. Smoking ≥5 cigarettes/day on average during 3 months prior to screening;
10. Pregnant or lactating women;
11. Positive pregnancy test before study drug administration, or male and female subjects who refuse to use effective contraceptive methods during and for 6 months post-trial, or who have plans to donate sperm or eggs;
12. Poor compliance or any other condition that in the investigator's opinion renders the subject unsuitable for trial participation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-03-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
(一) Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs). | Approximately 1 year
  Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs).

SECONDARY OUTCOMES:
PK(Pharmacokinetics):Tmax | Approximately 1 year
  Time to peak plasma concentration (Tmax)
PK(Pharmacokinetics):Cmax | Approximately 1 year
  Maximum serum concentration(Cmax)
PK(Pharmacokinetics):AUC | Approximately 1 year
  Area under the plasma concentration versus time curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China